CLINICAL TRIAL: NCT05394818
Title: An Open-label, Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Efficacy of SHR-A2009 for Injection in Patients With Advanced Solid Tumors
Brief Title: The Clinical Study of SHR-A2009 for Injection in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Suzhou Suncadia Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-A2009-I-102
Record Dates: First submitted 2022-05-24; First posted 2022-05-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-A2009 (Experimental)
  Interventions: Drug: SHR-A2009

INTERVENTIONS:
Drug: SHR-A2009 — The total dosage of SHR-A2009 was calculated according to the weight weighing results of the subjects before each administration, and was administered by intravenous drip.

SUMMARY:
This study is an open-label, phase I clinical trial of SHR-A2009 in patients with advanced solid tumors. The whole study is divided into three stages: dose escalation, dose expansion and efficacy expansion.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically or cytologically confirmed unresectable locally advanced or metastatic solid tumors which is relapsed or refractory to standard treatment, or lack of standard treatment, or standard treatment is not applicable currently;
2. Have at least one measurable tumor lesion per RECIST v1.1;
3. ECOG performance status of 0-1;
4. Life expectancy ≥ 12 weeks;
5. Adequate bone marrow and organ function.
6. Subjects must voluntarily agree to participate in the trial and sign a written informed consent form.

Exclusion Criteria:

1. Patients with active central nervous system metastases or meningeal metastases;
2. Ongoing or previous anti-tumor therapies within 4 weeks prior to the first dose of study drug;
3. Prior treatment with antibody-drug conjugate (ADC) consisting of topoisomerase I inhibitors;
4. History of serious cardiovascular and cerebrovascular diseases;
5. Severe infection within 4 weeks prior to the first dose;
6. Adverse reactions of previous anti-tumor treatment have not recovered to Grade ≤ 1 per NCI-CTCAE v5.0.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2022-07-21 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) or maximum administered dose (MAD) | From Day 1 to 90 days after last dose
  Incidence and category of dose limiting toxicities (DLTs) during the first cycle of SHR-A2009 treatment.
Recommended Phase 2 dose (RP2D) | From Day 1 to 90 days after last dose
  RP2D will be determined on the basis of evaluation on MTD/MAD, PK, efficacy data in dose escalation and dose expansion stages.
Incidence and severity of adverse events (AEs)/serious adverse events (SAEs) ([CTCAE] v5.0) | From Day 1 to 90 days after last dose
  Assess safety and tolerability of SHR-A2009 by way of adverse events (CTCAE v5.0).

SECONDARY OUTCOMES:
PK parameter: Tmax of SHR-A2009 | approximately 6 months
  Time to maximum concentration of SHR-A2009
PK parameter: Cmax of SHR-A2009 | approximately 6 months
  Maximum concentration of SHR-A2009
PK parameter: AUC0-t of SHR-A2009 | approximately 6 months
  area under the concentration-time curve from time 0 to the last measurable concentration time point of SHR-A2009
PK parameter: AUC0-∞ of SHR-A2009 | approximately 6 months
  area under the concentration-time curve from time 0 to infinity of SHR-A2009
Immunogenicity of SHR-A2009 | approximately 9 months
  Anti-SHR-A2009 antibody (ADA)
Overall response rate (ORR) | approximately within 36 months
  Evaluated using RECIST 1.1
Duration of response (DoR) | approximately within 36 months
  Evaluated using RECIST 1.1
Disease control rate (DCR) | approximately within 36 months
  Evaluated using RECIST 1.1
Progression-free survival (PFS) | approximately within 36 months
  Evaluated using RECIST 1.1

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital-Department of Medical Oncology, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided